CLINICAL TRIAL: NCT03379532
Title: Brain-computer Interface Controlled Neuromuscular Electrical Stimulation in Subacute Stroke
Brief Title: BCI-controlled NMES in Subacute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: Ecole Polytechnique Fédérale de Lausanne (Other); Clinique Romande de Readaptation (Network)
Responsible Party: Principal Investigator, Adrian Guggisberg, Médecin adjoint agrégé, assistant professor, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRSII5-170985B
Record Dates: First submitted 2017-12-14; First posted 2017-12-20 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- BCI-NMES (Active Comparator): Electrical stimulation of paretic upper limb is triggered contigent to voluntary motor cortex activation of the patient, as detected by the brain-computer interface.
  Interventions: Device: BCI-NMES
- Sham-NMES (Sham Comparator): Electrical stimulation of paretic upper limb is applied independently of motor cortex activation of the patient by using a prerecorded session of another patient.
  Interventions: Device: Sham-NMES

INTERVENTIONS:
Device: BCI-NMES — From the recorded brain activity (EEG) subject specific patterns will be extracted with machine learning techniques from recordings where the subject executes movements tasks. Whenever a subject-specific pattern can be identified and detected, this is used for triggering neuromuscular electrical stimulation.
  Arms: BCI-NMES
Device: Sham-NMES — Neuromuscular electrical stimulation is triggered independently of the patient's movement intentions.
  Arms: Sham-NMES

SUMMARY:
Stroke patients with severe upper limb movement deficits have limited treatment options and often remain severely handicapped at the chronic stage.

Recent findings have suggested that poor motor recovery can be due to severe damage of the cortico-spinal tract (CST), the neural fibres connecting the movement regions of the brain to the spinal cord. Hence, to improve recovery of upper limb movements it will be crucial to re-establish and strengthen CST projections.

Recent studies provided evidence that closed-loop brain computer interface-driven electrical stimulation of the paretic muscles can induce clinically important and lasting recovery of upper limb function, even in patients with chronic, severe motor affection. In this treatment approach, movement intentions of the patients are detected with electroencephalography and real-time analyses. This triggers an electrical stimulation of affected upper limb muscles.

In this study, the investigators hypothesize that neuromuscular electrical stimulation (NMES) applied contingent to voluntary activation of primary motor cortex, as detected by a brain-computer interface (BCI), can help restore CST projections. This might improve recovery of patients with severe upper limb movement deficits. Treatment will be started within the first 8 weeks after stroke onset.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke
* Stroke onset ≤ 8 weeks
* Severe, unilateral motor upper extremity hemiparesis (≤15 Fugl-Meyer Score)
* Ability to give informed consent

Exclusion Criteria:

* Second stroke during rehabilitation
* Skull breach
* Cardiac pacemaker
* Metallic implants in the brain
* Delirium or disturbed vigilance
* Inability to follow treatments sessions
* Severe language comprehension deficits
* Severe dystonia or spasticity
* Severe co-morbidity (ex, traumatic, rheumatologic, neurodegenerative diseases)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Upper Limb Fugl-Meyer Score, after treatment | Difference between the week before the intervention and the week after intervention
  Scale 0-66, higher scores indicate better outcome

SECONDARY OUTCOMES:
Change in motor evoked potential amplitude of the paretic arm | Difference between the week before the intervention and the week after intervention
  Continuous measure, higher amplitude changes indicate better outcome
Change in fractional anisotropy (FA) of the cortico-spinal tract as determined from diffusion tensor imaging | Difference between the week before the intervention and the week after intervention
  FA can have values between 0 and 1, higher values indicate better outcome
Change in electroencephalography functional connectivity | Difference between the week before the intervention and the week after intervention
  Computed from high-density EEG recordings. Continuous measure. Higher values indicate better outcome.

OTHER OUTCOMES:
Change in Upper Limb Fugl-Meyer Score, follow up | Difference between the week before intervention and 12 weeks after stroke onset
  Scale 0-66, higher scores indicate better outcome
Change in hand grip strength, after intervention | Difference between the week before the intervention and the week after intervention
  Jamar dynamometer. Continous measure expressed in kilograms. Higher values indicate better outcome.
Change in hand grip strength, follow up | Difference between the week before intervention and 12 weeks after stroke onset
  Jamar dynamometer. Continous measure expressed in kilograms. Higher values indicate better outcome.
Change in Functional Independence Measure (FIM) score, after intervention | Difference between the week before the intervention and the week after intervention
  Range 18-126, higher values indicate better outcome.
Change in Functional Independence Measure (FIM) score, follow up | Difference between the week before intervention and 12 weeks after stroke onset
  Range 18-126, higher values indicate better outcome.
Change in Semmes-Weinstein monofilament discrimination test, after intervention | Difference between the week before the intervention and the week after intervention
  Range 0.04 to 60 g. Lower values indicate better outcome.
Change in Semmes-Weinstein monofilament discrimination test, follow up | Difference between the week before intervention and 12 weeks after stroke onset
  Range 0.04 to 60 g. Lower values indicate better outcome.
Change in Modified Ashworth Score, after intervention | Difference between the week before the intervention and the week after intervention
  Range 0 to 4. Lower values indicate better outcome.
Change in Modified Ashworth Score, follow up | Difference between the week before intervention and 12 weeks after stroke onset
  Range 0 to 4. Lower values indicate better outcome.
Change in action research arm test (ARAT) score, after intervention | Difference between the week before the intervention and the week after intervention
  Scale range 0-57 points, higher values indicate better outcome.
Change in action research arm test (ARAT) score, follow up | Difference between the week before intervention and 12 weeks after stroke onset
  Scale range 0-57 points, higher values indicate better outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- University of Austin, Austin, Texas, United States
- Division of Neurorehabilitation, University Hospital of Geneva, Geneva, Canton of Geneva, Switzerland